CLINICAL TRIAL: NCT04893187
Title: A Phase 1 Study to Evaluate the Tolerance, Safety, Pharmacokinetics and Pharmacodynamics of Oral Administration of SSS17 in Chinese Healthy Adult Subjects With Single and Multiple Dose Escalation and the Effect of Food on the Pharmacokinetics of SSS17.
Brief Title: A Phase 1 Study of SSS17 in Healthy Subjects.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenyang Sunshine Pharmaceutical Co., LTD. (Industry)
Collaborators: Fifth Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SYSS-SSS17-UND-I-02
Record Dates: First submitted 2021-05-17; First posted 2021-05-19 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Anemia in Chronic Kidney Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Part 1: Single Dose Escalation SSS17 (Experimental): Escalating doses of SSS17, single dose administration
  Interventions: Drug: SSS17
- Part 1: Single Dose Escalation matching Placebo (Placebo Comparator): Escalating doses of matching placebo, single dose administration
  Interventions: Drug: Placebo
- Part 2: Multiple Dose Escalation SSS17 (Experimental): Escalating doses of SSS17, multiple dose administration
  Interventions: Drug: SSS17
- Part 2: Multiple Dose Escalation matching Placebo (Placebo Comparator): Escalating doses of matching placebo, multiple dose administration
  Interventions: Drug: Placebo
- Part 3: Treatment Sequence 1 (A to B) (Experimental): The subjects in the first cycle received oral administration of SSS17 on an empty stomach, and subjects in the second cycle received oral administration of SSS17 after a high-fat meal
  Interventions: Drug: SSS17
- Part 3: Treatment Sequence 2 (B to A) (Experimental): The subjects in the first cycle received oral administration of SSS17 after a high-fat meal, and the subjects in the second cycle received oral administration of SSS17 on an empty stomach
  Interventions: Drug: SSS17

INTERVENTIONS:
Drug: SSS17 — SSS17 is a novel small molecule compound which stimulates erythropoiesis through inhibition of hypoxiainducible factor- prolyl hydroxylases( HIF-PH). It is being developed for the treatment of anemia in patients with chronic kidney disease.
  Arms: Part 1: Single Dose Escalation SSS17; Part 2: Multiple Dose Escalation SSS17; Part 3: Treatment Sequence 1 (A to B); Part 3: Treatment Sequence 2 (B to A)
Drug: Placebo — Matched placebo.
  Arms: Part 1: Single Dose Escalation matching Placebo; Part 2: Multiple Dose Escalation matching Placebo

SUMMARY:
This study will investigate the efficacy, safety, pharmacokinetics and pharmacodynamics of single oral administration of 5 mg, 15 mg, 20 mg and 25 mg of SSS17 compared with placebo, and evaluate the efficacy, safety, tolerance, pharmacokinetics and pharmacodynamics of multiple oral administration of 15 mg and 20 mg of SSS17 compared with placebo. In addition, the study will assess the effect of food on the pharmacokinetics of SSS17.

DETAILED DESCRIPTION:
The study will enroll healthy volunteers from a single academic medical center in China. All participants will be informed about the study and potential risks and required to provide written informed consent prior to undergoing study-related procedures.The study will be divided into 3 parts.

Part 1: Subjects will be allocated 2:8 to receive placebo or SSS17（it was only 2:2 in 5mg dose group）,which will be administered by oral route with single dose. At each dose, tolerability, safety, PK and PD characteristics will be investigated.

Part 2: Subjects will be allocated 2:8 to receive placebo or SSS17, which will be administered by oral route with multiple dose. At each cohort，tolerability, safety, PK and PD characteristics will be investigated.

Part 3: The subjects will receive two cycles of treatment, one is given on an empty stomach, the other is given after a high-fat meal, with an interval of 15 days.

ELIGIBILITY:
Inclusion Criteria:

* Chinese healthy adult subjects aged 18-45 years (including the boundary value) at the time of signing the informed consent were male and female;
* In the screening period, the weight of male subjects was more than or equal to 50.0 kg; Female weight ≥ 45.0 kg; Body mass index (BMI) ranged from 19.0 kg / m2 to 26.0 kg / m2 (including boundary value); BMI = weight kg / height m2);
* Within 6 months from the date of signing the informed consent to the end of the trial, female subjects agreed to take reliable measures to avoid pregnancy and ensure no birth plan, while male subjects agreed to take reliable measures to avoid pregnancy and ensure no birth plan;
* Willing to participate in the study and sign a written informed consent, able to communicate well with the researchers, and agreed to follow the requirements of the trial protocol and follow-up on schedule.

Exclusion Criteria:

* Participated in other drug clinical trials within 3 months before screening;
* Have any clinical history of serious diseases or are suffering from related diseases, including but not limited to digestive system (such as diarrhea, vomiting, inflammatory bowel disease, hemorrhoids, acute gastritis, peptic ulcer, acute and chronic gastrointestinal disorders with obvious digestive and absorption disorders), cardiovascular system, respiratory system, urinary system, musculoskeletal system, endocrine system, gastrointestinal tract diseases, etc Diseases of nervous and mental system, blood system, immune system, etc; A history of any disease or thrombotic disease or vascular malformation that increases the risk of bleeding; Patients with dysphagia;
* Allergic constitution, known allergic to test drug ingredients or allergic history to any drug or food (mango, shrimp, crab, lobster, etc.) or pollen allergy history;
* Those who smoke more than 5 cigarettes / day or the same amount of tobacco after inquiry, or who can not ban smoking during the trial period; Or alcohol consumption per week is equal to 14 units (1 units 25mL wine Baijiu / 100mL wine / 285mL beer), or those who can not prohibit alcohol during the test period;
* Have a history of drug abuse or drug abuse;
* Within 6 months, there were fertility planning, sperm donation and egg donation planning;
* Patients with lactose intolerance (those who have had diarrhea after drinking milk);
* Those who have special requirements for diet and cannot accept unified diet;
* Blood donors or massive blood loss (≥ 400ml), EPO treatment, blood transfusion or use of blood products within 3 months before screening;
* Those vaccinated within 8 weeks before screening or during the study period;
* There was a history of acupuncture and blood sickness; Or with orthostatic hypotension;
* Those who have participated in and used the trial drug;Those who have used any prescription drug, over-the-counter drug, Chinese herbal medicine, vitamins or health care products within 14 days before screening and whose time is less than 5 half-life of the drug or less than 2 weeks (whichever is the longest);
* The serum pregnancy test of lactating and pregnant women, or female volunteers of childbearing age was positive;
* The results of physical examination, chest X-ray, color Doppler ultrasound, electrocardiogram and laboratory examination were abnormal and clinically significant; Or hemoglobin of male subjects was more than 175.0 g / L; Or hemoglobin of female subjects was more than 150.0 g / L; Or hemoglobin of male and female were less than 113g / L;
* Within 48 hours before enrollment, those who took any special diet that affected the absorption, distribution, metabolism and excretion of drugs, including pitaya, mango, grapefruit, lime, carambola or food or drink prepared from them, chocolate, and any food or drink containing caffeine;
* Urine drug screening test was positive;
* Alcohol breath test was positive within 24 hours before administration;
* The researchers think that there are other cases that are not suitable for the trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2021-07-26 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Part 1: AEs | Baseline up to Days 15
  Assessment AEs by frequency and severity in the part 1
Part 1: Maximum plasma concentration (Cmax) of SSS17 | Up to 336 hours post-dose
  Plasma samples will be collected and Cmax will be assessed in the part 1
Part 1: Area under the concentration-time curve (AUC) of plasma concentration of SSS17 | Up to 336 hours post-dose
  Plasma samples will be collected and the AUC from zero to infinity will be assessed in the part 1
Part 1: Time-to-Cmax (Tmax) of SSS 17 | Up to 336 hours post-dose
  Plasma samples will be collected and the Tmax will be assessed from the concentration-time curve in the part 1
Part 1: Elimination terminal half-life (t1/2) of SSS17 | Up to 336 hours post-dose
  Plasma samples will be collected and the t1/2 will be assessed in the part 1
Part 1: . Total amount of SSS17 excreted in urine over 72 hours (Ae0-72) | Up to 72 hours post-dose
  Urine sample will be collected at pre-specified intervals and Ae0-72 will be assessed in the part 1
Part 1: Fraction of SSS17 excretion during each collection interval (Fe0-72) | Up to 72 hours post-dose
  Urine sample will be collected at pre-specified intervals and Fe0-72 will be assessed in the part 1
Part 1: Renal clearance (CLR) of SSS17 | Up to 72 hours post-dose
  Urine sample will be collected at pre-specified intervals and CLR will be assessed in the part 1
Part 2: AEs | Up to Days 33 or 57
  Assessment AEs by frequency and severity in the part 2
Part 2: Steady state minimal concentration (Css_min) of SSS17 | Up to Days 33 or 57
  Plasma samples will be collected and Css_min will be assessed in the part 2
Part 2: Steady state maximum concentration (Css_max) of SSS17 | Up to Days 33 or 57
  Plasma samples will be collected and Css_max will be assessed in the part 2
Part 2: Steady state average concentration (Css_av) of SSS17 | Up to Days 33 or 57
  Plasma samples will be collected and Css_av will be assessed in the part 2
Part 2: Area under the concentration-time curve of plasma concentration of SSS17 within the interval of administration after reaching steady state (AUC0-τ) | Up to Days 33 or 57
  Plasma samples will be collected and the AUC from zero to τ will be assessed
Part 3: Maximum plasma concentration (Cmax) of SSS17 | Up to Days 44
  Plasma samples will be collected and Cmax will be assessed in the part 3
Part 3: Area under the concentration-time curve (AUC) of plasma concentration of SSS17 | Up to Days 44
  Plasma samples will be collected and the AUC from zero to infinity will be assessed in the part 3
Part 3: Time-to-Cmax (Tmax) of SSS 17 | Up to Days 44
  Plasma samples will be collected and the Tmax will be assessed from the concentration-time curve in the part 3
Part 3: Elimination terminal half-life (t1/2) of SSS17 | Up to Days 44
  Plasma samples will be collected and the t1/2 will be assessed in the part 3

SECONDARY OUTCOMES:
Part 1: EPO concentrations | Up to 168 hours post-dose
  Change of EPO concentrations from baseline following SSS17 in the part 1
Part 1: VEGF concentrations | Up to 168 hours post-dose
  Change of VEGF concentrations from baseline following SSS17 in the part 1
Part 1: Change of hepcidin from baseline | Up to 168 hours post-dose
  Change of serum hepcidin concentrations from baseline following SSS17 in the part 1
Part 1: Change of RTC from baseline | Baseline up to Days 15
  Change of RTC from baseline following SSS17 in the part 1
Part 1: Change of RBC from baseline | Baseline up to Days 15
  Change of RBC from baseline following SSS17 in the part 1
Part 1: Change of Hgb from baseline | Baseline up to Days 15
  Change of Hgb from baseline following SSS17 in the part 1
Part 2: EPO concentrations | Up to Days 33 or 57
  Change of EPO concentrations from baseline following SSS17 in the part 2
Part 2: VEGF concentrations | Up to Days 33 or 57
  Change of VEGF concentrations from baseline following SSS17 in the part 2
Part 2: Change of hepcidin from baseline | Up to Days 33 or 57
  Change of serum hepcidin concentrations from baseline following SSS17 in the part 2
Part 2: Change of RTC from baseline | Baseline up to Days 33 or 57
  Change of RTC from baseline following SSS17 in the part 2
Part 2: Change of RBC from baseline | Baseline up to Days 33 or 57
  Change of RBC from baseline following SSS17 in the part 2
Part 2: Change of Hgb from baseline | Baseline up to Days 33 or 57
  Change of Hgb from baseline following SSS17 in the part 2
Part 3: AEs | Up to Days 44
  Assessment AEs by frequency and severity in the part 3
Part 3: EPO concentrations | Up to Days 44
  Change of EPO concentrations from baseline following SSS17 in the part 3
Part 3: VEGF concentrations | Up to Days 44
  Change of VEGF concentrations from baseline following SSS17 in the part 3
Part 3: Change of hepcidin from baseline | Up to Days 44
  Change of serum hepcidin concentrations from baseline following SSS17 in the part 3
Part 3: Change of RTC from baseline | Baseline up to Days 44
  Change of RTC from baseline following SSS17 in the part 3
Part 3: Change of RBC from baseline | Baseline up to Days 44
  Change of RBC from baseline following SSS17 in the part 3
Part 3: Change of Hgb from baseline | Baseline up to Days 44
  Change of Hgb from baseline following SSS17 in the part 3

CONTACTS AND LOCATIONS:
Locations (1):
- The Fifth Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided